CLINICAL TRIAL: NCT04724174
Title: Double Purse-String Telescoped Pancreaticogastrostomy for High Risk Anastomosis: A 6-Year Single Center Case-Controlled Study
Brief Title: Pancreaticogastrostomy for High-Risk Pancreas
Acronym: GASTROPAN
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: GASTROPAN IPC-2020-029
Record Dates: First submitted 2021-01-19; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Anastomosis; Complications; Pancreatic Fistula
Keywords: High Risk Pancreatic Anastomosis; Clinically Relevant Pancreatic Fistula; Pancreaticogastrostomy
MeSH Terms: conditions — Pancreatic Fistula | interventions — Pancreaticojejunostomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreaticogastrostomy (PG) group: Patients underwent pancreatoduodenectomy with the PG technique
  Interventions: Procedure: pancreaticogastrostomy
- Pancreaticojejunostomy (PJ) group: Patients underwent pancreatoduodenectomy with the PJ technique
  Interventions: Procedure: pancreaticojejunostomy

INTERVENTIONS:
Procedure: pancreaticogastrostomy — Pancreaticogastrostomy technique was performed according to the precise description of Addeo et al.
  Groups: Pancreaticogastrostomy (PG) group
Procedure: pancreaticojejunostomy — Pancreaticojejunostomy technique was performed using the 5/0 polypropylene interrupted monofilament suture in a one-layered duct-to-mucosa end-to-side anastomosis (Cattell-Warren anastomosis).
  Groups: Pancreaticojejunostomy (PJ) group

SUMMARY:
In 2013, a double purse-string telescoped pancreaticogastrostomy (PG) technique appeared to significantly reduce the risk of postoperative pancreatic fistula (POPF). This study compared the incidence of clinically relevant POPF in patients with high-risk anastomosis after undergoing PG or pancreaticojejunostomy (PJ) techniques.

DETAILED DESCRIPTION:
From 2013 to 2019, consecutive patients with high-risk anastomosis (i.e., updated alternative-Fistula Risk Score (ua-FRS) >20%) underwent pancreatoduodenectomy with either the PJ or PG technique. Optimal mitigation strategy (external stenting and octreotide omission) was applied for all patients. The primary endpoint of the study was the incidence of clinically relevant POPF. Data were entered prospectively into an institutional clinical database (NCT02871336).

ELIGIBILITY:
Inclusion Criteria:

* Pancreatoduodenectomy
* High updated alternative -Fistula Risk Score which was defined > 20%, as the higher-risk category of the alternative-Fistula Risk Score

Exclusion Criteria:

* Explorative laparotomy
* Hard pancreatic parenchyma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with pancreatic tumor who underwent pancreatoduodenectomy
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically relevant post operative pancreatic fistula | at hospital discharge assessed up to 30 days
  clinically relevant post operative pancreatic fistula according to the 2016 International Study Group of Pancreatic Surgery (ISGPS) definition

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Turrini, PD, Principal Investigator — Institut Paoli-Calmettes- (IPC)

IPD SHARING:
Plan to Share IPD: No